CLINICAL TRIAL: NCT03741946
Title: The Effect of Contralateral Head Rotation on Internal Jugular Vein to Carotid Artery Distance and Overlap Ratio
Brief Title: Contralateral Head Rotation on Internal Jugular Vein to Carotid Artery Distance and Overlap Ratio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes025
Record Dates: First submitted 2018-11-07; First posted 2018-11-15 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Central Venous Catheterization; Surgery
Keywords: carotid arteries; central venous catheterization; jugular veins; Malay race; ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triangle of Sedillot identification using ultrasonography (Other): USG probe placed upright at the top of triangle of Sedillot at cricoid level
  Interventions: Procedure: Triangle of Sedillot identification using ultrasonography

INTERVENTIONS:
Procedure: Triangle of Sedillot identification using ultrasonography — Contralateral head rotation was done with protractor at angle 30°, 45°, and 60°. The distance and overlap ratio of IJV and CA was calculated in each angle.

SUMMARY:
This study aims to find out the effect of contra lateral head rotation to distance and overlapping of internal jugular vein and carotid artery at cricoid cartilage level by ultrasound guidance on the Malay race in Indonesia

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. 34 subjects were enrolled by using consecutive sampling method. Sample size was calculated by using numeric analytic comparative paired formula with repeated measurement. Inclusion criteria were patients with ASA score 1 and 2, aged between 18-60 years old, no anatomical abnormality in neck. Exclusion criteria were patients who were either obese, has history of previous central venous catheter cannulation, and limitation on contralateral head movement. Drop out criteria was abnormalities of anatomical IJV and CA. Basic demographic data, such as sex, age, body weight and height, body mass index were recorded. Patients were positioned in Trendelenburg (15°) position. Identification triangle of Sedillot at cricoid level in right neck with palpation at angle 0°. USG probe was placed upright at the top of triangle of Sedillot at cricoid level. Identification of IJV and CA was shown in transversal view then the IJV to CA distance and overlap ratio was calculated. Contralateral head rotation was done with protractor at angle 30°, 45°, and 60°. The distance and overlap ratio of IJV and CA was calculated in each angle.

ELIGIBILITY:
Inclusion Criteria:

* ASA score 1 and 2
* 18-60 years old
* no anatomical abnormality in neck

Exclusion Criteria:

* obese
* has history of previous central venous catheter cannulation
* limitation on contralateral head movement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
IJV to CA distance at different contralateral rotation angle | 2 months
  IJV to CA distance at different contralateral rotation angle (0°, 30°, 45°, 60°)
IJV to CA overlap ratio at different contralateral rotation angle | 2 months
  IJV to CA overlap ratio at different contralateral rotation angle (0°, 30°, 45°, 60°)

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lieberman JA, Williams KA, Rosenberg AL. Optimal head rotation for internal jugular vein cannulation when relying on external landmarks. Anesth Analg. 2004 Oct;99(4):982-988. doi: 10.1213/01.ANE.0000132908.77111.CA. PMID 15385337
- [Background] Troianos CA, Hartman GS, Glas KE, Skubas NJ, Eberhardt RT, Walker JD, Reeves ST; Councils on Intraoperative Echocardiography and Vascular Ultrasound of the American Society of Echocardiography. Guidelines for performing ultrasound guided vascular cannulation: recommendations of the American Society of Echocardiography and the Society of Cardiovascular Anesthesiologists. J Am Soc Echocardiogr. 2011 Dec;24(12):1291-318. doi: 10.1016/j.echo.2011.09.021. No abstract available. PMID 22115322
- [Background] Brass P, Hellmich M, Kolodziej L, Schick G, Smith AF. Ultrasound guidance versus anatomical landmarks for subclavian or femoral vein catheterization. Cochrane Database Syst Rev. 2015 Jan 9;1(1):CD011447. doi: 10.1002/14651858.CD011447. PMID 25575245
- [Background] Sibai AN, Loutfi E, Itani M, Baraka A. Ultrasound evaluation of the anatomical characteristics of the internal jugular vein and carotid artery--facilitation of internal jugular vein cannulation. Middle East J Anaesthesiol. 2008 Oct;19(6):1305-20. PMID 18942245
- [Background] Saitoh T, Satoh H, Kumazawa A, Nobuhara M, Machii M, Tanaka T, Shiraki K, Saotome M, Urushida T, Katoh H, Hayashi H. Ultrasound analysis of the relationship between right internal jugular vein and common carotid artery in the left head-rotation and head-flexion position. Heart Vessels. 2013 Sep;28(5):620-5. doi: 10.1007/s00380-012-0283-0. Epub 2012 Sep 12. PMID 22968853
- [Background] Troianos CA, Kuwik RJ, Pasqual JR, Lim AJ, Odasso DP. Internal jugular vein and carotid artery anatomic relation as determined by ultrasonography. Anesthesiology. 1996 Jul;85(1):43-8. doi: 10.1097/00000542-199607000-00007. PMID 8694381
- [Background] Miki I, Murata S, Nakazawa K, Onozawa S, Mine T, Ueda T, Yamaguchi H, Yasui D, Takeda M, Kumita S. Anatomical relationship between the common carotid artery and the internal jugular vein during head rotation. Ultrasound. 2014 May;22(2):99-103. doi: 10.1177/1742271X14524571. Epub 2014 Feb 25. PMID 27433202
- [Background] DeAngelis V, Denny J, Chyu D, Jan T, Lemaire A, Chiricolo A, Solina A. The Optimal Angle of Head Rotation for Internal Jugular Cannulation as Determined by Ultrasound Evaluation. J Cardiothorac Vasc Anesth. 2015 Oct;29(5):1257-60. doi: 10.1053/j.jvca.2015.02.007. Epub 2015 Feb 9. PMID 25998069
- [Background] Shoja MM, Ardalan MR, Tubbs RS, Loukas M, Vahedinia S, Jabbary R, Jalilvand M, Shakeri A. The relationship between the internal jugular vein and common carotid artery in the carotid sheath: the effects of age, gender and side. Ann Anat. 2008;190(4):339-43. doi: 10.1016/j.aanat.2008.04.002. Epub 2008 May 27. PMID 18595678